CLINICAL TRIAL: NCT06729645
Title: ACO/ARO/AIO-22 - External Beam Radiotherapy Combined with Endorectal High-dose-ratebrachytherapy in Elderly and Frail Patients with Rectal Cancer. a Prospective Multicentre Trial of the German Rectal Cancer Study Group
Brief Title: External Beam Radiotherapy Combined with Endorectal High-dose-rate Brachytherapy in Elderly and Frail Patients with Rectal Cancer
Acronym: ACO/ARO/AIO-22
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dr. Emmanouil Fokas, Prof Dr. med. Dr., University Hospital of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACO/ARO/AIO-22; 70115482 (Other Grant/Funding Number: German Cancer Aid (DKH))
Record Dates: First submitted 2024-11-27; First posted 2024-12-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Rectal cancer (Experimental): Patients will be initially treated with EBRT with 13 x 3 Gy to a total dose of 39 Gy to the primary tumor and pelvic lymph node, over a period of 2.5 weeks. Restaging with pelvic MRI and endoscopy will then be performed 6.5 weeks after completion of EBRT and prior to the first endorectal HDR-BT fraction to evaluate initial therapy response and the residual extent of the disease for target outlining. Following that, endorectal HDR-BT will be delivered with 3 x 8 Gy to a total dose of 24 Gy (dose prescription: 5 mm depth for cT1 tumors; 10 mm depth for cT2-3 tumors), with each endorectal brachytherapy application performed once weekly.
  Interventions: Other: radiotherapy

INTERVENTIONS:
Other: radiotherapy — External beam radiotherapy and endorectal brachytherapy

SUMMARY:
ACO/ARO/AIO-22 - External beam radiotherapy combined with endorectal high-dose-ratebrachytherapy in elderly and frail patients with rectal cancer.

A prospective multicentre trial of the German Rectal Cancer Study Group.

DETAILED DESCRIPTION:
Epidemiological data indicate that more than 50% of patients with newly-diagnosed rectal cancer are older than 70 years, with rising numbers expected over the next decades. Albeit total mesorectal excision (TME) is considered part of the standard multimodal therapy in rectal cancer, elderly and frail rectal cancer patients are often unable to undergo radical surgery as the risk of surgical complications and postoperative mortality rises with increasing age and comorbidity. In an analysis of the Colorectal Cooperative Group UK (1988-200) in 34.194 patients with colorectal cancer, 21% of those aged over 85 years did not undergo operation, while the rates of no surgical intervention were 11% in the 75-84 years age group. Furthermore, these patients often receive no treatment at all due to frailty and concurrent diseases, resulting in local and/or systemic disease progression with associated symptoms and impaired quality of life (QoL).

Significant advances have been made in modern radiotherapy (RT), which can provide a valuable alternative non-operative treatment strategy for elderly and frail patients. Notably, to achieve clinical complete response (cCR) with RT alone, high doses are needed. Recent data from randomized trials (OPERA, MORPEUS) in young and fit patients with rectal cancer indicate that increased RT doses can be safely delivered following external beam (chemo)radiotherapy (EBRT) followed by endoluminal radiotherapeutic modalities, such as contact X-ray brachytherapy (CXB) or high-dose rate endorectal brachytherapy (HDR-BT). However, prospective studies testing this therapeutic concept in elderly and frail patients with rectal cancer remain limited. Also, despite the wide availability of brachytherapy, applicability of this concept remains largely unexplored in this challenging age subgroup in Germany.

The ACO/ARO/AIO-22 prospective trial will aim to evaluate the efficacy of EBRT in combination with endorectal HDR-BT to achieve local control (cCR) and maintain QoL in elderly and frail patients with rectal cancer that are considered unfit for radical surgery, but amenable to EBRT in combination with endorectal HDR-BT or CXB.

The ACO/ARO/AIO-22 incorporates several aspects that make this prospective study important:

1. treatment decision making is challenging in elderly/frail patients with rectal cancer, whereas standardized treatment guidelines for this patient cohort are lacking, thus necessitating new clinical trials to establish the best possible treatment in this clinical setting;
2. the combination of EBRT and HDR-BT has been shown to result in high rates of tumor response with almost 90% overall response and cCR rates of approximately 50-80%, especially in young and fit patients with early stage tumors, whereas prospective trials in elderly/frail patients remain limited;
3. due to its very steep dose gradient, endorectal HDR-BT enables the delivery of a very high radiation dose to the tumor with a very steep decrease in the volume of normal tissue, thus increasing treatment efficacy while keeping toxicity low;
4. albeit already tested in different countries such as France, the Netherlands and the UK, the concept of combining EBRT with endorectal HDR-BT has not been widely tested in Germany yet and, thus, a prospective study is needed to evaluate its efficacy and safety in elderly/frail patients with rectal cancer, to develop expertise and to make this modality widely available for this challenging patient cohort.

Altogether, the concept of combining EBRT with endorectal HDR-BT to be tested as part of the ACO/ARO/AIO-22 prospective trial constitutes an attractive option in elderly/frail patients with rectal cancer unfit for radical surgery as it can potentially provide long-term local control of the primary tumor, prevent disease-related morbidity, prolong survival, improve QoL and even lead to cCR with complete cure in selected cases.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age ≥70 years) with a G8-frailty score ≤ 14 based on the G8 geriatric assessment tool of frailty and/or elderly patients (age ≥70 years) with American Society of Anesthesiologists Physical Status (ASA PS) ≥ 3 and/ elderly patients (age ≥70 years) unsuitable to tolerate radical surgery as judged by the surgeon and/or elderly patients (age ≥70 years) that refuse radical surgery
* Life expectancy ≥ 6 months
* Male and female patients with histologically confirmed diagnosis of rectal adenocarcinoma localized 0-16 cm from the anocutaneous line as measured by rigid rectoscopy
* MRI-defined cT1-3d N0/+ M0, mrCRM - / +, </= 2/3 involvement of the rectal wall circumference
* Staging requirements: High-resolution, thin-sliced (i.e. 3mm) magnetic resonance imaging (MRI) of the pelvis is the mandatory local staging procedure.
* Spiral-CT of the abdomen and chest to exclude distant metastases.

Exclusion Criteria:

* Previous or current drug abuse
* Other concomitant antineoplastic therapy
* Prior or concurrent malignancy ≤ 3 years prior to enrolment in study (Exception: non-melanoma skin cancer or cervical carcinoma FIGO stage 0-

  1), unless the patient is continuously disease-free
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Complete Response (cCR) or Near cCR at 12 Months | 12 Months
  The primary efficacy endpoint is the proportion of patients achieving a clinical complete response (cCR) or near cCR at 12 months after the initiation of treatment, assessed through MRI and endoscopic evaluation.
  Quality of Life (QoL) at 12 Months
  Assessed using the EORTC QLQ-ELD14 questionnaire, tailored to evaluate the QoL in elderly cancer patients. The primary measure will be the change in the QoL score from baseline to 12 months.

SECONDARY OUTCOMES:
Quality of Life and Functional Outcomes | 2 years
  EORTC QLQ-C30 and QLQ-CR29 for general and colorectal cancer-specific QoL. Wexner-Score for anorectal function assessment. Sustained cCR at 2 Years
  Proportion of patients maintaining a cCR for two years post-treatment. Disease-Free Survival (DFS) at 2 Years
  Time from treatment initiation to recurrence or death from any cause. Cumulative Incidence of Locoregional Regrowth
  Frequency of locoregional tumor regrowth in patients who initially achieved cCR.
  Cumulative Incidence of Distant Metastases Occurrence of distant metastases within the two-year follow-up period. Overall Survival (OS) at 2 Years Duration from treatment initiation to death from any cause. Acute and Late Toxicity Evaluation Categorized based on NCI CTCAE v.5.0, focusing on adverse events related to treatment.
  G8 Geriatric Assessment Evaluation of frailty and health status using the G8 assessment tool, both at baseline and during follow-ups.

OTHER OUTCOMES:
Translational/Biomarker Studies | 6 months
  Identification of molecular biomarkers predictive of treatment response or prognosis.
  Follow-Up Procedures Standardized Watch and Wait (W&W) protocol for patients achieving cCR or near cCR at six months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Fokas, MD DPhil, Study Chair — University Hospital of Cologne
Locations (4):
- Germany (4):
  - Klinikverbund Allgäu, Kempten, BaBaden-Württembergs
  - Frankfurt Universitätsklinikum, Frankfurt am Main, Hesse
  - Klinik für Strahlentherapie, Cyberknife und Radioonkologie Universität zu Köln, Cologne, North Rhine-Westphalia
  - Leipzig, Universitätsklinikum, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Access Criteria: ACO/ARO/AIO-22

REFERENCES:
- [Background] Fleischmann M, Diefenhardt M, Nicolas AM, Rodel F, Ghadimi M, Hofheinz RD, Greten FR, Rodel C, Fokas E; German Rectal Cancer Study Group. ACO/ARO/AIO-21 - Capecitabine-based chemoradiotherapy in combination with the IL-1 receptor antagonist anakinra for rectal cancer Patients: A phase I trial of the German rectal cancer study group. Clin Transl Radiat Oncol. 2022 Apr 6;34:99-106. doi: 10.1016/j.ctro.2022.04.003. eCollection 2022 May. PMID 35449546
- [Derived] Dapper H, Fleischmann M, Tselis N, Diefenhardt M, Hofheinz RD, Weiss C, Grabenbauer GG, Merten R, Grosu AL, Kirste S, Rieken S, Classen J, Langer C, Kuhnt T, Schmidberger H, Ghadimi M, Giordano F, Nestle U, Koerber SA, Bock F, Geiger M, Polat B, Bruns CJ, Dieplinger G, Popp F, Zander T, Brunner T, Tribius S, Arnold D, Wurschi G, Piso P, Friede T, Horner-Rieber J, Gkika E, Rodel C, Fokas E; German Rectal Cancer Study Group. ACO/ARO/AIO-22 - External beam radiotherapy combined with endorectal high-dose-rate brachytherapy in elderly and frail patients with rectal cancer: A prospective multicentre trial of the German Rectal Cancer Study Group. Clin Transl Radiat Oncol. 2025 Apr 13;53:100958. doi: 10.1016/j.ctro.2025.100958. eCollection 2025 Jul. PMID 40276115
- See also: Fleischmann, M., Dapper, H., Diefenhardt, M. et al. Perkutane Strahlentherapie kombiniert mit endorektaler Brachytherapie zum Organerhalt bei älteren/gebrechlichen Patienten mit Rektumkarzinom - die ACO/ARO/AIO-22-Studie. Onkologie 30, 129-132 (2024). ht — https://link.springer.com/article/10.1007/s00761-023-01470-2#Bib1